CLINICAL TRIAL: NCT05580484
Title: Efficacy and Safety of Purified Starch for Adhesion Prevention in Colorectal Surgery
Status: Completed | Type: Observational
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Tungcheng Chang, Chief of department of colorectal surgery, Taipei Medical University Shuang Ho Hospital
Other Study IDs: N202109018
Record Dates: First submitted 2022-10-09; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Adhesions Abdominal
MeSH Terms: interventions — Second-Look Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Purified starch/Control group: Patients who were willing to receive purified starch at their own expense during this first surgery were included in the purified starch group, and patients who did not re-ceive purified starch or other anti-adhesion products were included in the control group.
  Interventions: Procedure: Second surgery

INTERVENTIONS:
Procedure: Second surgery — The primary outcomes were adhesion severity and adhesion area in the lower ab-dominal cavity, as determined through direct visual observation of a laparotomy wound or laparoscopic observation from stoma closure wound.

SUMMARY:
Intra-abdominal adhesion occurs in up to 90% of patients after abdominal surgery. Many patient will undergo a second surgery for temporary stoma closure, therefore these ostomy closure operations can give an opportunity to evaluate adhesion caused by previous operations. This study was conducted to use second surgery to investigate the anti-adhesion effect of purified starch among patients who underwent colorectal surgery.

DETAILED DESCRIPTION:
Data was analyzed from the medical records of patients who underwent a second surgery after colectomy between January 2020 and April 2022. Patient were allocated to either the purified starch group and control group. Since January 2020, adhesion scores have been registered in operation note when patients undergo a second colorectal surgery. The primary outcomes in this study were adhesion severity and adhesion area. The secondary outcomes were operation time, blood loss, and postopera-tive complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent a second surgery after colorectal resection between January 2020 and April 2022 were enrolled into this study.

Exclusion Criteria:

* Patients who underwent a second surgery less than 1 month after the first colorectal resection or who developed peritoneum carcinomatosis in the second surgery and patients younger than 20 years were excluded.

Ages: 20 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent a second surgery after colorectal resection.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Adhesion severity | three to six months
  Adhesion severity was scored as grade 0 (no adhesion), grade I (filmy adhesion and blunt dissection), grade II (strong adhesion and sharp dissection), and grade III (very strong vascularized adhesion, sharp dissection, and damage barely preventable).
Adhesion area | three to six months
  Adhesion area was scored as grade 0 (no adhesion), grade I (adhesion of less than one-third of the area between the abdominal wall and the visceral organ in the lower abdominal cavity), grade II (adhesion of one-third and two-thirds of the area between the abdominal wall and the visceral organ in the lower abdominal cavity), and grade III (adhesion of more than two-thirds of the area between the abdominal wall and the visceral organ in the lower abdominal cavity).

CONTACTS AND LOCATIONS:
Overall Officials: Tung-Cheng Chang, Study Chair — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Taipei Medical University Shuang-Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided